CLINICAL TRIAL: NCT00800956
Title: An Open Label, Single Oral Dose Study to Investigate the Absorption, Metabolism and Excretion of [14C]-Esreboxetine.
Brief Title: Phase I Study to Determine the Absorption, Distribution, Metabolism and Excretion of Esreboxetine
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A6061018
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Radiolabel ADME study Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single oral dose of [14C]-esreboxetine (Experimental)
  Interventions: Drug: [14C]-esreboxetine

INTERVENTIONS:
Drug: [14C]-esreboxetine — Single oral dose of 6mg esreboxetine in solution containing approximately 100uCi [14C]-esreboxetine

SUMMARY:
The purpose of the study is to learn more about how esreboxetine is handled by the body i.e. the absorption, metabolism and excretion of esreboxetine.

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects aged 45 to 65 years Body mass index (BMI=weight/height2) 18 to 30 kg/m2

Exclusion Criteria:

Any clinically relevant abnormality identified on the screening medical assessment Any condition possibly affecting drug absorption Subjects with exposure to significant radiation (eg serial Xray or CT scans, barium meal etc)or who have participated in a radiolabelled study in the past 12 months, or who have occupational exposure to radioactivity History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5ounces (150ml) of wine or 12 ounces (360ml) of beer or 1.5 ounces (45ml) of hard liquor) within 6 months of screening 12-lead ECG demonstrating QTc>450mses at screening Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of radioactivity in urine and and faeces as a percentage of the total radioactive dose administered over time. Collection of plasma, urine and faeces for the assessment of parent drug and metabolites of esreboxetine where possible | Approx 10 days
Pharmacokinetic parameters of esreboxetine and identification and abundance of metabolites in plasma, urine and faeces if possible | Approx 10 days

SECONDARY OUTCOMES:
Clinical safety data | Approx 10 days
Pharmacokinetic parameters of plasma esreboxetine metabolites if possible | Approx 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061018&StudyName=Phase%20I%20study%20to%20determine%20the%20absorption%2C%20distribution%2C%20metabolism%20and%20excretion%20of%20esreboxetine